CLINICAL TRIAL: NCT05626452
Title: Implementation and Dissemination of Evidence-Based Interventions to Improve PrEP Care Continuum Outcomes Among Women in Community Health Clinics in the Southern U.S.
Brief Title: PrEP Optimization Among Women to Enhance Retention and Uptake
Acronym: POWER Up
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: AllianceChicago (Other); Howard Brown Health Center (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Northwestern University (Other); Rush University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB21-0971
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: PrEP Uptake
Keywords: Pre-exposure prophylaxis; Stepped-wedge randomized trial

STUDY DESIGN:
Intervention Model Description: This study will use a cluster randomized, cross-sectional stepped wedge study with 12 clusters (8 CHCs from the South and 4 CHCs from the Midwest) to evaluate the effect of the intervention package as compared to the control condition (usual care) on the proportion of PrEP prescriptions among eligible participants. Cross-sectional data from participants who are eligible for PrEP will be collected at 6 different calendar intervals of 6 months ("steps"). Although all clusters will begin the study in the control condition (usual care), beginning in step 3 at each six-month interval three randomly chosen CHCs (containing a mix of Southern and Midwestern CHCs) will switch from the control condition to the intervention condition. Beginning at step 2, the step prior to 3 CHCs switching from control to intervention condition will be spent in a six-month transition period. This design will allow for data collection at all CHCs to contain observations from both intervention and control periods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): The current mechanisms used at each healthcare site to assess HIV risk/ take a sexual history, assess PrEP eligibility, identify PrEP ineligibility for otherwise PrEP eligible patients, provide PrEP education, offer PrEP, provide PrEP navigation, measure PrEP uptake, and measure PrEP persistence/retention.
- Intervention (Experimental): Implementation of 1) Patient Education, 2) Provider PrEP training, 3) EMR optimization, and 4) PrEP navigation, and the effect of these intervention components on the ability of each site to assess HIV risk/take a sexual history, assess PrEP eligibility, identify PrEP ineligibility for otherwise PrEP-eligible patients, provide PrEP education, offer PrEP, provide PrEP navigation, measure PrEP uptake, and measure PrEP persistence/retention.
  Interventions: Behavioral: PrEP Education; Behavioral: Provider training; Other: EMR Optimization; Other: PrEP Navigation; Other: Provider Audit and Feedback

INTERVENTIONS:
Behavioral: PrEP Education — Education for participants regarding PrEP
  Arms: Intervention
Behavioral: Provider training — Training for medical providers at CHCs about how to identify participants eligible for PrEP, how to perform behavioral risk assessment and discussion of PrEP, and how to prescribe PrEP and monitor PrEP
  Arms: Intervention
Other: EMR Optimization — EMR modifications to enhance PrEP care continuum outcomes including HIV risk assessment, identification of participants eligible for PrEP, provision of PrEP education, clinical decision support tools for prescription of PrEP, and tracking of PrEP care continuum outcomes using an electronic population health management tool
  Arms: Intervention
Other: PrEP Navigation — Use of CHC staff members to assist participants with obtaining PrEP and attending PrEP care appointments
  Arms: Intervention
Other: Provider Audit and Feedback — Audit of provider rates of PrEP prescription and persistence among participants and regular provision of feedback to providers with their performance on these PrEP measures
  Arms: Intervention

SUMMARY:
Black women experience one of the highest incidences of HIV among all subpopulations in the United States, but pre-exposure prophylaxis (PrEP) use among Black cisgender women is very limited. The investigators will implement four strategies (provider training, patient education, EMR optimization, and PrEP navigation) at 12 community health clinics in the Midwest and South. The investigators predict that PrEP use and other related outcomes will improve for participants after the intervention period.

DETAILED DESCRIPTION:
Research Design After the investigators have adapted the POWER-Up strategies for use in the new setting, the investigators will conduct a hybrid type II trial within the framework of a cluster randomized, cross-sectional stepped wedge study. The investigators will use the RE-AIM framework for evaluation. The investigators will utilize a cluster randomized, cross-sectional stepped wedge trial, including sites in the South and the Midwest. This study design will allow us to roll out the intervention across diverse geographic areas and assess the change in clinical and implementation outcomes from the pre-intervention (control) and the post intervention (intervention) periods. The cluster, or unit of analysis, is each CHC, N=12 (8 in the South, 4 in the Midwest). In a stepped wedge study, each cluster contributes both time and observations to the control condition (usual care) and the intervention condition (strategies to increase PrEP use). Every cluster switches from the control to the intervention at regular time intervals ("steps"), but at different points in calendar time. More than one cluster may start the intervention at a step, but the step at which a cluster switches from control to intervention is randomized. The design is cross-sectional as outcomes are obtained from the subset of patients seen during each time period at each clinic rather than following individually recruited patients over time. This use of clinics under both intervention and control conditions improves precision when intra-cluster correlation is high, which is likely among the CHCs the investigators have chosen.

In our stepped wedge design, each step is 6 months long, and there are 4 waves of intervention implementation (three sites begin the intervention at the same step, a mix from the South and the Midwest, N=12). Three CHC sites will be randomized to each step occurring at 6-month intervals. Each cluster also undergoes a 6-month transition period when the individual clinics will prepare to implement the intervention package.

Although the investigators hypothesize that the effect of this intervention will increase PrEP uptake among participants, the investigators powered this study to ensure that the investigators could detect a range of intervention effectiveness. The investigators used the R statistical package swCRTdesign V3.1 to verify that a sample of 50 participants at 6 different times ("steps") each lasting 6 months, at the 12 CHC sites ("clusters") provides adequate power (>80%) to detect a change from a baseline of 1% of eligible participants receiving prescriptions for PrEP to 2% with an ICC of 0.2 and a CAC of 0.80.60. This minimum sample size per time interval is one that can easily be met by all of the clinics used as sites in this study (100 eligible participants per calendar year).

A key element of the research infrastructure will be AllianceChicago's uniform EMR system, which is distinguished by the integration of evidence-based practice recommendations into the end user interface to provide clinical decision support at the point of care. AllianceChicago's information technology (IT) team will create a study specific fields to measure study outcomes. The IT team will build custom reports in their data warehouse to access and validate in real-time. Reports will be built to pull data (ICD, CPT/HCPCS, and RXNORM codes, laboratory results, demographic characteristics) from the medical record and billing claims, and will be used to determine implementation success for the RE-AIM outcomes of effectiveness and maintenance. The investigators will utilize the Health Catalyst Tool which already has reports built to monitor PrEP care continuum outcomes. Additional reports will be built to monitor: 1) Participants who receive HIV risk assessment 2) participants who receive PrEP education; 3) participants who receive PrEP navigation; 4) PrEP prescriptions among eligible participants.

Implementation Patient education: CHC staff will perform HIV risk assessment for participants who present at the CHCs for care. HIV risk assessment will consist of asking questions regarding PrEP indications adapted from the USHS guidelines for PrEP (e.g., sexual partners, recent STIs, condom use, drug use, etc). For participants who meet criteria of "PrEP eligibility," patient education regarding PrEP will be provided. Patient education occurs at each clinic visit.

Provider training: Providers will complete 3 sessions of 1-hour virtual trainings regarding PrEP (providing patient education, identifying PrEP-eligible participants, offering PrEP, etc.). CHCs will provide protected time for providers to complete the trainings. Trainings will be virtual but also interactive, including the opportunities for providers to use electronic avatars to practice difficult conversations with virtual participants. Monthly audit and feedback will be provided post-training to measure and support sustained behavior change. The investigators will integrate PrEP outcomes reports into the overall quality metric reporting for each clinic. Every month the medical director of each clinic reviews quality metrics for the clinical site. The medical director reports the metrics during monthly clinic meetings and steps are taken to address any metrics that fall short of the expected benchmark. Data on clinic staff's use of PrEP clinical decision support tools and PrEP care continuum outcomes will be incorporated into standard monthly quality report. During monthly site check-ins, the investigators will review this data with the medical director and clinical champions.

EMR optimization: AllianceChicago will incorporate PrEP clinical decision support, including PrEP indication documentation, PrEP order set, and electronic notifications of PrEP-eligible participants into the CHC's EMR and provide weekly reports of PrEP care continuum outcomes for the CHC to review and act upon.

PrEP navigation: The investigators will work with the CHCs to engage staff in the adapted PrEP support roles using manualized procedures and training. PrEP navigators will meet with participants 2-3 times initially to support PrEP uptake, and will check in with patients monthly thereafter (appointment, refill reminders will be based on participants' own schedules).

Monitoring and Process Evaluation with Feedback: The investigators will track the implementation process and provide feedback and support to the CHC for challenges in implementing the strategies, as well as ongoing feedback on interim outcomes including number of participants who underwent HIV risk assessment, the number who discussed PrEP with a provider, proportion initiating PrEP, and results of provider training. Results will be discussed between the research team and each CHC to understand barriers and identify and document adaptations needed using Stirman's FRAME methodology. Broadly, the investigators will discuss and document (1) what and why the investigators adapted, (2) goals of the adaptation, (3) who was involved in the adaptation process, (4) when the investigators adapted, (5) forms of adaptation, and (6) measurement and evaluation.

Evaluation: Utilizing the RE-AIM framework, the investigators will evaluate the success of the implementation strategies. The investigators will gather feedback from CHC providers, staff, and participants using mixed methods with both quantitative surveys and qualitative interviews. For evaluation of the provider training, The investigators will use the Kirkpatrick four-level training evaluation model. The investigators will use provider-level quantitative surveys to assess the four-levels of training: satisfaction and perceived value (Level 1); knowledge and self-efficacy (Level 2); application of knowledge (Level 3; i.e., number of participants offered PrEP); and effectiveness (Level 4; i.e., the increase in proportion of participants on PrEP). Data regarding number of participants who had PrEP education, discussions, and who initiated and persisted on PrEP will be collected from the EMR with electronic reports developed by AllianceChicago. To assess provider and CHC staff feedback about the implementation strategies, the investigators will use surveys to assess the following measures: Acceptability of Intervention Measure (AIM)), appropriateness (Intervention Appropriateness Measure (IAM)), and feasibility (Feasibility of Intervention Measure (FIM)). In addition, the investigators will recruit 400 participants to complete surveys regarding acceptability (AIM) of the POWER Up strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* HIV-negative

Exclusion Criteria:

* Younger than age 18 years
* HIV-positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
PrEP uptake | Baseline through 36 months
  Number of participants initiating PrEP

SECONDARY OUTCOMES:
PrEP persistence consecutive months | Baseline through 36 months
  Number of participants with six consecutive months of PrEP prescriptions
PrEP persistence amount of coverage | Baseline through 36 months
  Number of participants who achieve appropriate coverage of PrEP (Coverage in days required: 154/180 (per six months))
HIV risk assessment PrEP ineligibility | Baseline through 36 months
  Number of participants who undergo HIV risk assessment
PrEP eligibility | Baseline through 36 months
  Number of participants identified as PrEP eligible
PrEP ineligibility | Baseline through 36 months
  Number of participants identified as PrEP ineligible
PrEP offered | Baseline through 36 months
  Number of participants offered PrEP
PrEP navigation | Baseliend through 36 months
  Number of participants receiving PrEP navigation services
PrEP Education | Baseline through 36 months
  Number of participants receiving PrEP education
Eligibility for PrEP Education | Baseline through 36 months
  Number of participants who meet the following criteria: Age >18, do not have HIV, are attending an appointment where PrEP could be prescribed
Provider feedback | Baseline through 36 months
  Number of CHC providers receiving feedback regarding their PrEP prescription rates
Change in provider knowledge and attitudes about PrEP | Baseline through 36 months
  Average change in score between baseline and post intervention quiz on provider knowledge and attitudes about PrEP
Change in patient knowledge and attitudes about PrEP | Post-intervention, month 37
  Average change in score between baseline and post intervention quiz on patient knowledge and attitudes about PrEP
Provider training | Post-intervention, month 37
  Number of providers who complete online training
Providers who educate patients about PrEP | Baseline through 36 months
  Number of providers who offer PrEP education to participants
Provider prescription of PrEP | Baseline through 36 months
  Number of providers who prescribe PrEP to participants
Acceptability for providers | Post-intervention, month 37
  Average score among providers of the Acceptability of Intervention Measure tool (AIM)
Acceptability for patients | Post-intervention, month 37
  Average score among patients of the Acceptability of Intervention Measure tool (AIM)
Appropriateness | Post-intervention, month 37
  Average score among providers of the Intervention Appropriateness Measure tool (IAM)
Appropriateness | Post-intervention, month 37
  Average score among patients Intervention Appropriateness Measure tool (IAM)
Maintenance | Post-intervention, month 37
  Average score among providers of the Program Sustainability Assessment Tool (PSAT)
Feasibility of intervention | Post-intervention, month 37
  Average score among providers on the Feasibility of Intervention Measure tool (FIM)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Ridgway, MD, MS, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Devlin SA, Ridgway JP, Dawdani A, Enaholo OE, Liegeon G, Kasal N, Pyra M, Hirschhorn LR, Simon J, Haider S, Ducheny K, Johnson AK. Adapting Provider Training and Pre-Exposure Prophylaxis Advertising to Increase Pre-Exposure Prophylaxis Awareness and Uptake Among Black Cisgender Women. AIDS Patient Care STDS. 2023 Dec;37(12):574-582. doi: 10.1089/apc.2023.0188. Epub 2023 Nov 21. PMID 38011350